CLINICAL TRIAL: NCT03767491
Title: Smartphone Cognitive Behavioral Therapy for Obsessive-Compulsive Disorder: A Randomized, Waitlist-control Trial
Brief Title: Waitlist-Control Trial of Smartphone CBT for Obsessive-Compulsive Disorder (OCD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study must be registered under the sponsor instead of the site, so we have created a new posting in the sponsor's account.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Telefónica S.A. (Industry)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Chief of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018P001669-a
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2020-05

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Smartphone-delivered CBT for OCD (Experimental): 12-week Smartphone delivered CBT for OCD.
  Interventions: Device: Smartphone-delivered CBT for OCD
- 12 Week Waitlist Control (Other): 12-week waitlist control. (Note: participants will be crossed over to 12-week Smartphone-delivered CBT for OCD following the 12-week waitlist control).
  Interventions: Device: Smartphone-delivered CBT for OCD

INTERVENTIONS:
Device: Smartphone-delivered CBT for OCD — 12-week Smartphone-delivered CBT for OCD. In-person cognitive-behavioral therapy (CBT) is an empirically supported treatment for OCD. The app-delivered CBT in this project includes modules such as cognitive skills (e.g., cognitive restructuring, core belief work), behavioral skills (e.g., exposure with ritual prevention), and perceptual retraining/mindfulness skills.

SUMMARY:
The investigators are testing the efficacy of Smartphone-delivered cognitive behavioral therapy (CBT) treatment for obsessive compulsive disorder (OCD). The investigators hypothesize that participants receiving app-CBT will have greater improvement in Y-BOCS scores than those in the waitlist condition at treatment endpoint (week 12).

DETAILED DESCRIPTION:
The primary aims of this study are to test the efficacy of a Smartphone-based CBT treatment for adults with OCD recruited nationally. Eligible subjects (N=58) will be randomly assigned to 12 weeks of Smartphone-delivered CBT for OCD either immediately, or after a 12-week long waiting period (50-50 chance). The investigators hypothesize that Smartphone-delivered CBT for OCD will be feasible and acceptable to individuals with OCD, and that it will lead to greater reductions in OCD symptom severity compared to the passage of time (waitlist control).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* current diagnosis of primary DSM-5 OCD, based on MINI
* currently living in the United States

Exclusion Criteria:

* Psychotropic medication changes within 2 months prior to enrollment (Participants taking psychotropic medication must have been on a stable dose for at least 2 months prior to enrollment and not change medication during study period)
* Past participation in ≥ 4 sessions of CBT for OCD
* Current severe substance use disorder
* Lifetime bipolar disorder or psychosis
* Acute, active suicidal ideation as indicated by clinical judgment and/or a score ≥ 2 on the suicidal ideation subscale of the C-SSRS
* Current severe comorbid major depression, as indicated by clinical judgment and/or a QIDS-SR total score ≥ 21
* Concurrent psychological treatment
* Does not own a supported mobile Smartphone with a data plan
* Lack of technology literacy that would interfere with ability to engage with smartphone treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Difference in OCD severity (Y-BOCS) at the end of treatment/waitlist period. | Endpoint (week 12)
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is the gold-standard, semi-structured clinician-administered assessment of OCD severity. It contains 10 items ranging from 0 to 4, which are summed to generate a total score (range = 0-40). Higher scores indicate more severe OCD symptoms. The Y-BOCS will be used to assess change in OCD symptoms from baseline to endpoint.

SECONDARY OUTCOMES:
Difference in depression at the end of treatment/waitlist period | Endpoint (week 12)
  Participants who receive app-CBT will have greater improvement on depression (QIDS-SR). The QIDS-SR is a self-report measure of depressive symptoms consisting of 16 scale items with responses ranging from 0 to 3, including one suicide item (item #12). Higher scores correspond with greater depression severity, and the measure is a well-validated, sensitive measure of symptom severity in depression.
Difference in functional impairment at the end of treatment/waitlist period | Endpoint (week 12)
  Participants who receive app-CBT will have greater improvement on functional impairment (SDS). The SDS uses a Likert scale from 0 (not at all) to 10 (extremely) to assess impairment in occupational, social, and family domains. Higher scores indicate greater impairment.
Difference in quality of life at the end of treatment/waitlist period | Endpoint (week 12)
  Participants who receive app-CBT will have greater improvement on quality of life, assessed using The Quality of Life, Enjoyment, and Satisfaction Questionnaire - Short Form (Q-LES-Q). The Q-LES-Q-SF is a self-report measure of subjective quality of life, containing Likert items ranging from 1 (Very Poor) to 5 (Very Good). Total scores are presented as a percentage of the maximum value (i.e., ranging from 0 to 100, with higher scores indicating greater quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Anna Schwartzberg, Boston, Massachusetts, United States